CLINICAL TRIAL: NCT02733965
Title: Impact of Clinical Pharmacy Consultations in Patients With Cancer Treated With Oral Anti-cancer Therapies on the Rate of Serious Adverse Events
Acronym: PharmaOnco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-03
Record Dates: First submitted 2016-03-22; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Oral Anticancer Therapy.
Keywords: clinical pharmacy consultations; oral anti-cancer therapy; serious adverse events; medication reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard course (Other): The patients in the control group will have a "classic" course of treatment. They will receive -An educational assessment consisting on evaluating the patient's educational needs.
  * Group workshops entitled "Disease and drugs", "Dietary and sports activity", "Psychology Workshop" during which the patient will be able to participate in order to get all the information he needs.
  * Individual therapeutic education sessions to specifically and personally highlight certain non-pharmaceutical educational needs identified at the time of the educational assessment.
  Moreover, in the control arm, a systematic "short pharmaceutical interview" with an average duration of 15 minutes will be proposed to patients at the initiation of treatment, at D15 after the prescription (considered as the date of inclusion) at M1 and then every 3 months (M3, M6, M9 and M12):
  Interventions: Other: No Pharmaceutical Consultations
- Long Pharmaceutical Consultations (Other): The patients will receive the same course of treatment as in the control group, including the D0 short pharmaceutical interview, with the same prerogatives of acceptance or rejection of participation in the TPE program. Short pharmaceutical interviews from D15 to M12 will be replaced by long pharmaceutical consultations of 30 to 60 minutes. The latter consisting in a full clinical medication review and incorporating the pedagogic aspects addressed in the short pharmaceutical interviews but for all therapeutic drugs taken by the patient. Additional consultations are possible on the request of the oncologist and/or patient. The consultations carried out at the request of the oncologist and/or the patient will be counted The first part of the pharmaceutical consultation focuses on a complete clinical medication review including Establishment of the patient profile: medical history, drug allergies and intolerance, comorbidities, age, understanding capacities, organizational capacity
  Interventions: Other: Pharmaceutical Consultations

INTERVENTIONS:
Other: Pharmaceutical Consultations — The first part of the pharmaceutical consultation focuses on a complete clinical medication review, the effective use of drugs will be discussed with the patient.
  Study of health behaviors Concerning self-medication and alternative medicine Addictions Drug adherence List and grade (NCI version 4) of clinical signs and laboratory abnormalities The biological data will be obtained Clinical signs will be obtained from patient questioning The second part of the consultation is to achieve firstly a pharmaco-therapeutic analysis of the treatment in order to detect problems with drugs as classified by the French Society of Clinical Pharmacy The third step consists on providing "pharmaceutical interventions" following the pharmaco-therapeutic analysis (18).
  These pharmaceutical interventions might concern the prescribers, the other caregivers, or the patient himself. T
  Arms: Long Pharmaceutical Consultations
Other: No Pharmaceutical Consultations
  Arms: standard course

SUMMARY:
The improvement of the care pathway of oncology patients through Clinical Pharmacy activities for outpatients (such as pharmaceutical consultation) should be implemented and evaluated.

In order to improve the care pathway of patients on anticancer oral therapies, The investigators suggest in this research project to integrate into the medical care a "Clinical Pharmacy follow-up" for the patient at the hospital in the form of "pharmaceutical consultations". These pharmaceutical consultations carried out in coordination with the hospital clinical teams also aim to make the link between the hospital and community pharmacists.

DETAILED DESCRIPTION:
The improvement of the care pathway of oncology patients through Clinical Pharmacy activities for outpatients (such as pharmaceutical consultation) should be implemented and evaluated.

In order to improve the care pathway of patients on anticancer oral therapies, the investigators suggest in this research project to integrate into the medical care a "Clinical Pharmacy follow-up" for the patient at the hospital in the form of "pharmaceutical consultations". These pharmaceutical consultations carried out in coordination with the hospital clinical teams also aim to make the link between the hospital and community pharmacists. These pharmaceutical consultations were initiated in Marseille and Grenoble University Hospitals in order to know the special needs of patients under oral chemotherapies. However, the impact of these pharmaceutical consultations in a population of patients receiving ambulatory oral therapy remains unknown and needs to be evaluated using objective criteria such as the rate of adverse events which the consequences are considerable both for the patient and the society.

These observations prompted us to establish a randomized controlled study with the objective of assessing the impact of the Clinical Pharmacy consultations in cancer patients treated with oral anti-cancer therapies on the general care management: occurrence of serious adverse events (primary outcome).

This bicenter, prospective, randomized, placebo-controlled, open-label, two-parallel group study is performed to assess the efficacy of pharmaceutical consultations in the experimental group (full clinical medication review) and pharmaceutical interviews in the control group (Patient Therapeutic Education for oral anticancer drugs only). Depending on the result of the randomization the patient will find himself in one of those 2 parallel arms:

* Control group: standard course + short pharmaceutical interviews (therapeutic education)
* Experimental group: standard course + long pharmaceutical consultations (including full clinical medication review and therapeutic education)

Control group: therapeutic education through short pharmaceutical interviews

The patients allocated in the control group will have a "classic" course of treatment. They will receive the best medical care and will be offered to participate in the therapeutic education program in place in the participating centers including:

* An educational assessment consisting on evaluating the patient's educational needs.
* Group workshops entitled "Disease and drugs", "Dietary and sports activity", "Psychology Workshop" during which the patient will be able to participate in order to get all the information he needs.
* Individual therapeutic education sessions to specifically and personally highlight certain non-pharmaceutical educational needs identified at the time of the educational assessment.

Moreover, in the control arm, a systematic "short pharmaceutical interview" with an average duration of 15 minutes will be proposed to patients at the initiation of treatment, at D15 after the prescription (considered as the date of inclusion) at M1 and then every 3 months (M3, M6, M9 and M12):

* Dosage, including the maximum dosage for modular taken drugs
* Duration of treatment
* User precautions
* The necessary information to drug use
* Any special precautions to be taken and any information relevant to the good understanding of the treatment by the patient
* Biological analyzes necessary for the initiation, monitoring, and pursuit of certain treatments

Experimental group: Clinical Pharmacy through Long Pharmaceutical Consultations In this experimental group, patients will receive the same course of treatment as the patients in the control group, including the D0 short pharmaceutical interview, with the same prerogatives of acceptance or rejection of participation in the TPE program. Short pharmaceutical interviews from D15 to M12 will be replaced by long pharmaceutical consultations of 30 to 60 minutes. The latter consisting in a full clinical medication review and incorporating the pedagogic aspects addressed in the short pharmaceutical interviews but for all therapeutic drugs taken by the patient. Additional consultations are possible on the request of the oncologist and/or patient. The consultations carried out at the request of the oncologist and/or the patient will be counted.

The first part of the pharmaceutical consultation focuses on a complete clinical medication review including:

* Establishment of the patient profile: medical history, drug allergies and intolerance, comorbidities, age, understanding capacities, organizational capacity…
* Establishment of the list of current treatments (cancer treatment, treatment of comorbidities, self-medication, other products). The effective use of drugs will be discussed with the patient.
* Study of health behaviors:

  * Concerning self-medication (reasons, active ingredients, doses, etc.) and alternative medicine
  * Addictions (smoking, alcohol...)
  * Drug adherence
* List and grade (NCI version 4) of clinical signs and laboratory abnormalities:

  * The biological data will be obtained on the basis of biological test results addressed to the oncologist and all other test results provided by the patient
  * Clinical signs will be obtained from patient questioning The second part of the consultation is to achieve firstly a pharmaco-therapeutic analysis of the treatment (level 3 pharmaceutical analysis according to the criteria of the French Society of Clinical Pharmacy) in order to detect problems with drugs as classified by the French Society of Clinical Pharmacy (18).

The third step of the consultation consists on providing "pharmaceutical interventions" following the pharmaco-therapeutic analysis (18).

These pharmaceutical interventions might concern the prescribers, the other caregivers, or the patient himself. These interventions will be done in the absolute respect for the French Code of Public Health. All these interventions will be documented, tracked, and evaluated, particularly in terms of acceptance by prescribers.

Sample size Both centers have the necessary number of patients needed to ensure the proper recruitment required for the study.

The annual throughput of the AP-HM is about 300 patients. Targeted diseases as part of this research project are gastrointestinal tumors (GIST, colorectal), neuroendocrine, renal, gynecological, urological (prostate) and skin (melanoma) cancers. The annual throughput of Grenoble University Hospital is more than 70 patients. Targeted diseases are renal tumors, breast and colorectal cancers.

The number of subjects to be included required is determined from the primary endpoint, namely the rate of adverse events of grade III-IV. Data from the current practice in the main center (AP- HM) and from the literature estimate this rate at 35%.

The majority of adverse events related to drugs being preventable, the investigators estimate a decrease of 20 points in this rate in the experimental arm, that is to say a rate of 15%. 166 subjects (83 per group) are needed for a power of 90% and an alpha risk of 5%. To compensate the potential lost of the out of sights (estimated around 15%), the investigators will include 190 subjects in total.

The sample size was determined to obtain 90% power to detect a 20 percent difference in between the 2 groups, as this difference is considered to be clinically significant. In accordance with previous studies (26-31), the investigators hypothesized that the occurrence of the primary endpoint will be at 35% in the control group. With the threshold for statistical significance set at a p-value of 0.05 (two-sided alpha), these calculations showed that 166 patients are needed (83 per group). Assuming that potentially 15% of patients will be lost to follow-up, a total of 190 individuals need to be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of both sexes
* Patients with cancer pathology whatever stage/grade and associated comorbidities he has
* Patients treated with oral cancer therapy for less than a month regardless of the therapy line
* Have accepted to participate and signed the non-opposition form

Exclusion Criteria:

* Patients less than 18 years of age and all vulnerable people, in accordance with French laws (pregnant women, adults under guardianship or trusteeship; persons deprived of liberty)
* Patients under treatment for more than one month
* Patients refusing to participate in the research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Rate of grade III-IV adverse events defined by the NCI criteria | 6 months

SECONDARY OUTCOMES:
Adverse events by the NCI criteria | 1st, 3rd, 6th, 9th, 12th months of the study
Satisfaction toward the treatment: satisfaction with medicines questionnaire ((SatMed-Q®) | 1st, 3rd, 6th, 9th, 12th months of the study
The number of visit to the emergency services | 1st, 3rd, 6th, 9th, 12th months of the study
The number of hospitalizations | 1st, 3rd, 6th, 9th, 12th months of the study
The number of additional medical consultations | 1st, 3rd, 6th, 9th, 12th months of the study
Drug adherence: Morisky scale 8-item; | 1st, 3rd, 6th, 9th, 12th months of the study
Quality of life: Short Form 36 (SF-36) questionnaire | 1st, 3rd, 6th, 9th, 12th months of the study
Survival: RECIST criteria | 1st, 3rd, 6th, 9th, 12th months of the study

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No